CLINICAL TRIAL: NCT05286814
Title: Phase II Study Evaluating the Efficacy of PDS01ADC in Combination With Hepatic Artery Infusion Pump (HAIP) and Systemic Therapy for Subjects With Metastatic Colorectal Cancer, Intrahepatic Cholangiocarcinoma, or Metastatic Adrenocortical Carcinoma
Brief Title: PDS01ADC in Combination With Hepatic Artery Infusion Pump (HAIP) and Systemic Therapy for Subjects With Metastatic Colorectal Cancer, Intrahepatic Cholangiocarcinoma, or Metastatic Adrenocortical Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10000307; 000307-C
Record Dates: First submitted 2022-03-12; First posted 2022-03-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01-22

CONDITIONS: Metastatic Colorectal Cancer (Mcrc); Intrahepatic Cholangiocarcinoma (Icc); Intrahepatic Bile Duct Cancer; Colorectal Neoplasms; Colorectal Cancer; Cholangiocarcinoma; Bile Duct Neoplasms; Bile Duct Cancer; Adrenocortical Carcinoma (ACC); Adrenal Cortical Carcinoma; Adrenal Gland Cancer; Adrenal Gland Neoplasms; Adrenal Cortex Neoplasms
Keywords: Unresectable Liver Tumor; SMART System; Response Rates; Progression Free Survival (Pfs); Patient Survival; Overall Survival (Os); NHS-IL12; Mcrc; Icc; ACC
MeSH Terms: conditions — Colorectal Neoplasms; Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension; Bile Duct Neoplasms; Adrenocortical Carcinoma; Adrenal Gland Neoplasms; Adrenal Cortex Neoplasms | interventions — Dexamethasone; Floxuridine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/ HAIP +PDS01ADC+FOLFOX or FOLFORI (Experimental): PDS01ADC+HAIP FUDR and Dexamethasone chemotherapy in combination with FOLFOX or FOLFIRI
  Interventions: Drug: Dexamethasone; Drug: PDS01ADC; Device: Intera 3000 Hepatic Artery Infusion Pump (HAIP); Drug: Floxuridine
- 2/ HAIP +PDS01ADC+GemOx or FOLFOX (Experimental): PDS01ADC+HAIP FUDR and Dexamethasone chemotherapy in combination with GemOx or FOLFOX
  Interventions: Drug: Dexamethasone; Drug: PDS01ADC; Device: Intera 3000 Hepatic Artery Infusion Pump (HAIP); Drug: Floxuridine
- 3/ HAIP +PDS01ADC+GemOx (Experimental): PDS01ADC+HAIP FUDR and Dexamethasone chemotherapy in combination with GemOx
  Interventions: Drug: Dexamethasone; Drug: PDS01ADC; Device: Intera 3000 Hepatic Artery Infusion Pump (HAIP); Drug: Floxuridine

INTERVENTIONS:
Drug: Dexamethasone — HAIP FUDR and Dexamethasone treatment on D1 of every cycle. Dexamethasone: (1 mg/day X pump volume / pump flow rate)
Drug: PDS01ADC — PDS01ADC will be administered by subcutaneous injection on Day 15 of every cycle. Cycle 1 at 12 mcg/kg; Cycle 2 reduced to 8 mcg/kg with the addition of systemic chemotherapy, to continue for further cycles. Note: any dose reduction in FUDR = 50% due to liver enzyme elevations means that the dose of PDS01ADC will be reduced to 4 mcg/kg.
Device: Intera 3000 Hepatic Artery Infusion Pump (HAIP) — Intera 3000 HAIP will be filled with mixture of Floxuridine and Dexamethasone in 25,000 units heparin/saline (Heparin + 0.9% Sodium Chloride) on Day 1; Days 1-14 of every cycle pump will perfuse drugs to liver. On Day 15 of each cycle, the pump will be emptied and filled with 30,000 units heparin/saline (Heparin + 0.9% Sodium Chloride); Days 15-28 of every cycle will perfuse heparin/saline to liver.
Drug: Floxuridine — HAIP FUDR and Dexamethasone treatment on D1 of every cycle. Floxuridine: (0.12 mg/kg x ideal average body weight in kg X 30 mL [pump volume] / Pump Flow Rate)

SUMMARY:
Background:

One way to treat liver cancer is to deliver chemotherapy drugs only to the liver (and not to the whole body). Researchers want to see if adding the drug PDS01ADC can improve the treatment. The drug triggers the immune system to fight cancer.<TAB>

Objective:

To see if treatment with HAIPs to deliver liver-directed FUDR and Dexamethasone chemotherapy in combination with PDS01ADC is effective for certain cancers.

Eligibility:

People aged 18 and older who have cancer of the bile ducts that is only in the liver, or colorectal cancer that has spread to the liver, or cancer of the adrenal glands that has spread to the liver, who are also receiving or planning to receive standard systemic chemotherapy for their disease.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood tests

Pregnancy test (if needed)

Tumor biopsy (if needed)

Electrocardiogram

Computed tomography (CT) scans

Participants will have an abdominal operation. A catheter will be placed into an artery that feeds blood to the liver. The catheter will then be attached to the HAIP. The HAIP will lay under the skin on the left side of the abdomen.

All participants will have liver-directed FUDR and Dexamethasone chemotherapy drugs or heparin with saline infused into the HAIP every 2 weeks. PDS01ADC will be injected under the skin every 4 weeks. They will receive this treatment until their cancer gets worse or they have bad side effects.

Participants will also receive standard systemic chemotherapy for their disease, assigned based on diagnosis, through an IV by their medical oncologist (at NIH or by a local provider) every 2 weeks.

Participants will have 2 study visits at NIH each month. They will have CT scans every 8 weeks. At visits, they will repeat some screening tests.

Participants will have a follow-up visit 1 month after treatment ends. Then they will be contacted every 6 months for 5 years.

DETAILED DESCRIPTION:
Background:

Regional chemotherapy for hepatic malignancies takes advantage of the fact that tumors are perfused almost exclusively by the hepatic artery and, that the agent used (Floxuridine, FUDR) has a 95% first-pass metabolism by the liver.

Early clinical trials performed during the 1970's and 1980's demonstrated impressive response rates that led to the adoption of hepatic artery infusion pump chemotherapy (HAIP) at select centers; however, little has changed in the ensuing decades with respect to regional

therapy for the liver, although there has been continued and even renewed interest.

Dose reductions of FUDR are common after several treatments, which has limited both the magnitude and duration of treatment responses in many cases.

We posit that the logical and much-needed "next step" in regional therapy is to take advantage of the FUDR-induced tumor necrosis with an agent able to activate local tumor immunity for a synergistic effect.

PDS01ADC is an immunocytokine composed of two IL-12 heterodimers, each fused to the H-chain of the NHS76 antibody. The NHS76 IgG1 antibody has affinity for both single- and double-stranded DNA (dsDNA), and targets regions of tumor necrosis where DNA has become exposed. PDS01ADC targets necrotic areas of the tumor and activates immune cells in the tumor microenvironment to induce a Th1 polarization of lymphocytes and the release of IFN-gamma. IFN-gamma in turn induces a host of immunomodulatory effects that contribute to robust antitumor responses that are localized within the tumor microenvironment, with no systemic distribution or exposure to IL-12.

Data from a recent Phase I study demonstrate that subcutaneous administration of PDS01ADC is safe and a MTD has been determined. Moreover, preclinical models indicate that PDS01ADC synergizes with therapies able to effectively induce tumor necrosis, which may also minimize toxicity by limiting off-target exposure.

Objective:

-To determine the objective response rate (ORR) in participants with unresectable metastatic colorectal cancer (mCRC), intrahepatic cholangiocarcinoma (ICC), or adrenocortical carcinoma (ACC) with liver dominant disease treated with PDS01ADC in combination with HAIP in participants receiving systemic therapy

Eligibility:

* Histologically or cytologically confirmed, unresectable, colorectal adenocarcinoma metastatic to the liver (Cohort 1), intrahepatic cholangiocarcinoma (Cohort 2) or adrenocortical carcinoma with liver dominant disease (Cohort 3)
* No evidence of extrahepatic metastases
* Participants must have received first-line systemic chemotherapy.
* Age >= 18 years

Design:

-Open label, single center, non-randomized Phase II study

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria- All Cohorts

* Participants must have a documented diagnosis of one of the following cancers:

  * Metastatic colorectal cancer (mCRC)
  * Intrahepatic cholangiocarcinoma (ICC)
  * Adrenocortical carcinoma (ACC) with liver dominant disease
* Participants must have an identified medical oncologist who has recommended and is planning to oversee treatment with one of the following standard chemotherapy regimens (based on disease type) not to begin sooner than 28 days after initiation of study-directed HAIP intervention:

  * mCRC: FOLFOX or FOLFIRI
  * ICC: GemOx or FOLFOX
  * ACC: GemOx
* Age >= 18 years.
* Negative serum or urine pregnancy test at screening for individuals of childbearing potential (IOCBP).

NOTE: IOCBP is defined as any individual who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal. IOCBP must have a negative pregnancy test (HCG blood or urine) during screening.

* All participants (regardless of childbearing potential) must agree to use highly effective contraception prior to study entry, for the duration of study participation, and for 3 months after completion of study treatment for those able to father a child or 6 months after completion of study treatment for those of child-bearing potential (i.e., IOCBP). Highly effective birth control (failure rate of less than 1%), e.g., intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner and sexual abstinence. Note: The use of condoms by participants who are able to get other individuals pregnant is required unless the partner of childbearing potential is permanently sterile.
* Nursing (including breastfeeding) participants must agree to discontinue nursing.
* Arterial anatomy on CT angiogram or CT chest, abdomen and pelvis multiphase (i.e., CT C/A/P multiphase) amenable to placement of the HAIP.
* Participant must sign the informed consent form to participate in this study.
* HIV-positive participants may be considered for this study only if they have an undetectable viral load.
* Participants must agree to co-enroll on the Surgical Oncology Program s tissue collection protocol 13C0176, "Tumor, Normal Tissue and Specimens from Patients Undergoing Evaluation or Surgical Resection of Solid Tumors".
* Participant's liver metastases must not be amenable to resection/ablation to No Evidence of Disease (NED) in one stage.

Inclusion Criteria-Metastatic Colorectal Carcinoma

* Participants must have histologically or cytologically confirmed diagnosis of colorectal adenocarcinoma metastatic to the liver (Cohort 1).
* Participants must have measurable liver metastatic disease.
* Participants must have received 1st line systemic chemotherapy.
* ECOG performance status <= 1.
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes > 3,000/mcL
  * absolute neutrophil count > 1,500/mcL
  * platelets > 90,000/mcL
  * hemoglobin > 8 g/dL
  * total bilirubin < 1.5 X institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR eGFR within normal as predicted by the CKD-EPI equation > 60 mL/min/1.73 m2.

Inclusion Criteria-Intrahepatic Cholangiocarcinoma

* Participants must have histologically or cytologically confirmed diagnosis of intrahepatic cholangiocarcinoma confined to the liver (Cohort 2). Archival tumor sample may be used but if archival tissue is not available or is not adequate, tissue biopsy will be required.
* Clinical or radiographic evidence of metastatic disease to regional (porta hepatis) lymph nodes will be allowed, provided it is amenable to resection.
* Participants must have radiographically measurable disease.
* Disease must be considered unresectable at the time of preoperative evaluation.
* Participants must have received 1st line systemic chemotherapy.
* ECOG performance status <=1.
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes >= 2,000/ mm^3
  * absolute neutrophil count > 1,500/mcL
  * platelets >= 75,000/ mm^3
  * hemoglobin > 8 g/dL
  * total bilirubin < 1.5 mg/dl
  * creatinine <= 1.5 mg/dl

Inclusion Criteria-Adrenocortical Carcinoma

* Participants must have histologically or cytologically confirmed diagnosis of adrenocortical carcinoma (ACC), also referred to as "adrenocortical cancer".
* Participants must have received at least one line of systemic chemotherapy.
* Participants must have measurable liver metastatic disease.
* ECOG performance status <= 1.
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes > 3,000/mcL
  * absolute neutrophil count > 1,500/mcL
  * platelets > 90,000/mcL
  * hemoglobin > 8 g/dL
  * total bilirubin < 1.5 X institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) < 3 X institutional upper limit of normal
  * creatinine < 2 X institutional upper limit of normal

EXCLUSION CRITERIA:

Exclusion Criteria- All Cohorts

Participants who are receiving any other investigational agents.

* Participants who have previously received rIL-12.
* Participants with active autoimmune diseases, that might deteriorate when receiving an immunostimulatory agent with the exceptions:

  * diabetes type I, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible;
  * participants requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses <= 10 mg of prednisone or equivalent per day;
  * administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is eligible.
* History of organ transplant, except for transplants that do not require immunosuppression.
* History of or active inflammatory bowel disease (e.g., Crohn s disease, ulcerative colitis).
* Known hypersensitivity or allergic reactions attributed to any compounds of similar chemical or biologic composition to the study medication, such as recombinant IL-12 or other monoclonal antibodies and history of allergic reactions attributed to compounds of similar chemical composition to FUDR or heparin.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke < 6 months prior to enrollment, myocardial infarction < 6 months prior to enrollment, unstable angina, congestive heart failure (>= NYHA III) or serious cardiac arrhythmia requiring medication.
* All conditions associated with significant necrosis of nontumor-bearing tissues.
* Esophageal or gastroduodenal ulcers < 6 months prior to treatment.
* Active ischemic bowel disease.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Active concurrent malignancies within the last five years other than colorectal primary except basal cell skin carcinoma and thyroid carcinoma.
* Prior radiation to liver.
* Participants with active Hepatitis B or C infection.
* Significant acute or chronic infections (i.e., tuberculosis) history of exposure or history of positive tuberculosis test; plus, presence of clinical symptoms, physical or radiographic findings).
* Any condition, including the presence of laboratory abnormalities and/or insufficient normal liver parenchyma, which places the participant at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study.

Exclusion Criteria-Metastatic Colorectal Carcinoma

-Participants with incontrovertible radiographic evidence of disease outside of the colon/rectum (primary) and liver given unlikelihood of benefit from liver-directed therapy.

Note: Lung lesions seen on CT do not always represent metastases. They are very hard to qualify, therefore exception to this exclusion is participants with fewer than five lung lesions greater than 1 cm that have not increased in size by more than 10% over a 4-month period of time and are amenable to resection should subsequent problematic growth occur. Lesions less than 1 cm are indeterminant as far as etiology is concerned and will be ignored. Participants with liver metastases and oligometastatic lung lesions (we define oligometastatic as less than 5 amenable to thoracoscopic removal) are still likely to benefit from liver directed therapy.

* Participants who have undergone extra-hepatic metastasectomy and have a documented disease-free interval less than or equal to 4 months.
* Participants with a history of MSI-high results who need to be treated with check-point inhibitors.
* Prior treatment with FUDR.

Exclusion Criteria-Intrahepatic Cholangiocarcinoma

-Presence of distant metastatic disease. Clinical or radiographic evidence of metastatic disease to regional lymph nodes will be allowed, provided it is amenable to resection.

Note: Lung lesions seen on CT do not always represent metastases. They are very hard to qualify, therefore exception to this exclusion is participants with fewer than five lung lesions greater than 1 cm that have not increased in size by more than 10% over a 4-month period of time and are amenable to resection should subsequent problematic growth occur. Lesions less than 1 cm are indeterminate as far as etiology is concerned and will be ignored. Participants with liver metastases and oligometastatic lung lesions (we define oligometastatic as less than 5 amenable to thoracoscopic removal) are still likely to benefit from liver directed therapy.

* Prior treatment with FUDR.
* Diagnosis of sclerosing cholangitis.
* Clinical evidence or portal hypertension (ascites, gastroesophageal varices, or portal vein thrombosis).

Exclusion Criteria-Adrenocortical Carcinoma

* Participants with incontrovertible radiographic evidence of additional abdominal disease outside of the liver (including the primary tumor) that is not amenable to complete surgical extirpation at the time of pump placement.
* Clinical evidence or portal hypertension (ascites, gastroesophageal varices, or portal vein thrombosis).
* Diagnosis of sclerosing cholangitis.
* Participants with pulmonary metastases that have progressed by RECIST criteria in the preceding 3 months prior to study enrollment.
* Participants with known mismatch repair mutation who have not been treated with a checkpoint inhibitor. Acceptable methods of MSI testing for history of MSI results include immunohistochemistry (IHC) and next generation sequencing (NGS) of tumor material.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine overall response rates | baseline, every 8 weeks while on treatment, and 4-8 weeks following initial documentation of objective response; an additional scan is performed at Week 12.
  Simon optimal two-stage Phase II trial design will be used to determine overall response using RECIST criteria. The clinical response rate (CR+PR) will be determined and reported along with a 95% confidence interval, separately by cohort.

SECONDARY OUTCOMES:
Determine overall survival (OS) | date of enrollment until death from any cause, or after 5 years off treatment
  CT will be used for response criteria. Overall survival (OS) probability will be determined using Kaplan-Meier estimates for all participants, separately by cohort; the median OS will be reported along with a 95% confidence interval.
Determine extra-hepatic progression-free survival (PFS) | date of operation to date of first observation of progressive disease within the liver or death, or after 5 years off treatment whichever comes first
  CT will be used for response criteria. Extra-hepatic progression-free survival (PFS) probability will be determined using Kaplan-Meier estimates for all participants, separately by cohort; the median PFS will be reported along with a 95% confidence interval.
Evaluate safety of PDS01ADC in combination with HAIP therapy | on-going from treatment start through end of treatment visit
  Safety will be assessed by analyzing the type, grade and frequency. Toxicities by grade and per participant will be determined and reported separately by disease cohort.
Determine hepatic progression-free survival (PFS) | date of operation to date of first observation of progressive disease within the liver or death, or after 5 years off treatment whichever comes first
  CT will be used for response criteria. Hepatic progression-free survival (PFS) probability will be determined using Kaplan-Meier estimates for all participants, separately by cohort; the median PFS will be reported along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Hernandez, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Victory JH, Smith EC, Ryan CE, Lambdin J, Sarvestani AL, Friedman LR, Eade AV, Larrain C, Pu T, Luberice K, Ramamoorthy B, Rainey AJ, Hannah CE, Smith KM, Mabry D, Xie C, Davis JL, Blakely AM, Gulley JL, Schlom J, Monge C, Greten TF, Hernandez JM. Hepatic artery infusion pump (HAIP) therapy in combination with targeted delivery of IL-12 for patients with metastatic colorectal cancer or intrahepatic cholangiocarcinoma: a phase II trial protocol. J Gastrointest Oncol. 2024 Jun 30;15(3):1348-1354. doi: 10.21037/jgo-24-71. Epub 2024 Jun 20. PMID 38989414
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000307-C.html